CLINICAL TRIAL: NCT00168116
Title: To Evaluate the Effects of Transfer of Submandibular Salivary Gland to the Submental Region (Outside the Radiation Field) on Xerostomia in Head and Neck Cancer Patients Receiving Radiation as the Primary Treatment Versus Patients Who Will Not Have Such a Procedure
Brief Title: Xerostomia in Head and Neck Cancer Patients Receiving Radiation as the Primary Treatment Versus Patients Who Will Not Have Such a Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16620
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Head and Neck Cancer
Keywords: nasopharynx; xerostomia; prevention
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia | interventions — Radiotherapy; Surgical Procedures, Operative; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: radiation treatment and surgery
Procedure: radiation alone

SUMMARY:
The purpose of this study is to compare the side effects of radiation treatment and surgery versus radiation alone, where no surgery is done to move the salivary gland and place it under the chin region where it can be shielded from radiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological diagnosis of squamous cell carcinoma
* Patients with unilateral or no neck involvement of the nasopharynx
* The submandibular transfer will be done on the uninvolved side of the neck.
* Karnofsky score greater than or equal to 70
* Expected survival greater than one year
* A signed informed consent

Exclusion Criteria:

* Bilateral neck nodes involvement. Involvement of level 1 lymph nodes on the side of the proposed procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2000-07; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Quality of life

SECONDARY OUTCOMES:
Treatment interruptions
Incidence of percutaneous endoscopic gastronomy (PEG)
Incidence of oral candidiasis
Overall survival
Disease free survival
Pattern of recurrence
Complications

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Jha, MBBA, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada